CLINICAL TRIAL: NCT06028464
Title: The Effect of Multiple Doses of Carbamazepine on the Pharmacokinetics of a Single Oral Dose of BI 1810631 in Healthy Male Subjects (an Open-label, Two-period, Fixed-sequence Trial)
Brief Title: A Study in Healthy Men to Test Whether Carbamazepine Influences the Amount of Zongertinib in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1479-0011; 2022-503046-50-00 (Other: CTIS)
Record Dates: First submitted 2023-08-30; First posted 2023-09-08 (Actual); Results first posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Healthy
MeSH Terms: interventions — Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zongertinib Alone (Reference)/ Zongertinib+Carbamazepine (Test) (Experimental): Participants took a single 60 mg oral dose of Zongertinib after fasting overnight (reference period). In the test period, they took the same Zongertinib dose after 18 days of daily Carbamazepine pretreatment, with doses increasing from 200 mg to 600 mg. They continued taking 600 mg of Carbamazepine daily for 6 days after the Zongertinib dose.
  Interventions: Drug: Zongertinib; Drug: Carbamazepine

INTERVENTIONS:
Drug: Zongertinib — Participants were administered a single dose of 60 milligrams (mg) of Zongertinib film-coated tablet orally on Day 1 with 240 milliliters (mL) of water after an overnight fast of at least 10 hours.
  Other Names: Hernexeos®
Drug: Carbamazepine — Participants received increasing doses of Carbamazepine once daily as extended-release tablets with 240 mL of water for 18 days, starting at 200 mg, then 400 mg, and finally 600 mg. Afterward, they continued taking 600 mg of Carbamazepine once daily for 6 days.

SUMMARY:
The main objective of this trial is to investigate the effect of multiple oral doses of the strong CYP3A inducer carbamazepine on the pharmacokinetics of a single dose of BI 1810631 in plasma.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG, the neurological examination, or the skin inspection) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Further exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was an open-label, two-treatment, two-period, fixed-sequence crossover trial in healthy male Participants comparing the test treatment (T) with the reference treatment (R). Treatment R consisted of one single oral dose of 60 mg zongertinib as a film-coated tablet alone. Treatment T consisted of one single oral dose of 60 mg zongertinib as a film-coated tablet with multiple oral doses of carbamazepine, titrated from 200 mg once daily (q.d.) to 400 mg q.d., then to 600 mg q.d.
Pre-assignment Details: A total of 16 participants entered the trial after being screened for eligibility, ensuring they met all inclusion and none of the exclusion criteria. They were allocated to the same treatment sequence to receive 2 treatments in a fixed order (R-T). All 16 received the first treatment (R), and 15 received the second (T). One participant did not start the second treatment due to a positive drug test result but completed the follow-up visit and was not considered to have prematurely discontinued.
Groups:
- Zongertinib Alone (Reference)/ Zongertinib+Carbamazepine (Test): Zongertinib Alone:
  In the reference treatment period, participants were administered a single dose of 60 milligrams (mg) of Zongertinib film-coated tablet orally on Day 1 with 240 milliliters (mL) of water after an overnight fast of at least 10 hours.
  Zongertinib + Carbamazepine:
  In the test treatment period (Period 2), participants were administered a single oral dose of 60 milligrams (mg) of Zongertinib in tablet form after an overnight fast of at least 10 hours, with 240 milliliters (mL) of water. This followed 18 days of pretreatment with increasing doses of Carbamazepine, starting at 200 mg, then 400 mg, and finally 600 mg, administered once daily as extended-release tablets with 240 mL of water. Additionally, subjects continued to receive 600 mg of Carbamazepine once daily for 6 days following Zongertinib administration.
Period: Period 1: Reference Treatment Period (R)
Arm/Group | Zongertinib Alone (Reference)/ Zongertinib+Carbamazepine (Test)
Started | 16
Completed | 16
Not Completed | 0
Period: Washout
Arm/Group | Zongertinib Alone (Reference)/ Zongertinib+Carbamazepine (Test)
Started | 16
Completed | 15
Not Completed | 1
Not completed — Positive drug test. | 1
Period: Period 2: Test Treatment Period (T)
Arm/Group | Zongertinib Alone (Reference)/ Zongertinib+Carbamazepine (Test)
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set includes all participants who were treated with at least one dose of trial drug.
Arm/Group | Zongertinib Alone (Reference)/ Zongertinib+Carbamazepine (Test)
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.5 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Zongertinib in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of Zongertinib in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
  Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model.
Time Frame: One hour before administration of zongertinib, and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 11, 12, 24, 36, 48, 72, 120, and 168 hours after administration.
Population: Pharmacokinetic parameter analysis set (PKS): This set includes all participants in the treated set (TS) who provided at least one PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Standard Error); unit: hour * nanomole / liter (h*nmol/L)
Groups:
- Zongertinib Alone (Reference, R): In the reference treatment period (Period 1), participants were administered a single oral dose of 60 milligrams (mg) of Zongertinib in tablet form following an overnight fast of at least 10 hours, with 240 milliliters (mL) of water.
- Zongertinib+Carbamazepine (Test, T): In the test treatment period (Period 2), participants were administered a single oral dose of 60 milligrams (mg) of Zongertinib in tablet form after an overnight fast of at least 10 hours, with 240 milliliters (mL) of water. This followed 18 days of pretreatment with increasing doses of Carbamazepine, starting at 200 mg, then 400 mg, and finally 600 mg, administered once daily as extended-release tablets with 240 mL of water. Additionally, subjects continued to receive 600 mg of Carbamazepine once daily for 6 days following Zongertinib administration.
Arm/Group | Zongertinib Alone (Reference, R) | Zongertinib+Carbamazepine (Test, T)
Number analyzed (Participants) | 16 | 15
hour * nanomole / liter (h*nmol/L) | 12334.87 (NA) — Adjusted geometric standard error = 1.06 | 4500.05 (NA) — Adjusted geometric standard error = 1.06
Statistical Analysis 1: Comparison: Zongertinib Alone (Reference, R) vs Zongertinib+Carbamazepine (Test, T); Ratio of adjusted geometric means was calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model; Test type: Other; Adjusted geometric mean ratio (%) = 36.48, 90% CI 2-sided [31.96 to 41.64] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 21.9

2. Primary Outcome: Maximum Measured Concentration of Zongertinib in Plasma (Cmax)
Description: Maximum measured concentration of Zongertinib in plasma (Cmax). Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: nanomole / liter (nmol/L)
Arm/Group | Zongertinib Alone (Reference, R) | Zongertinib+Carbamazepine (Test, T)
Number analyzed (Participants) | 16 | 15
nanomole / liter (nmol/L) | 914.01 (NA) — Adjusted geometric standard error = 1.10 | 515.84 (NA) — Adjusted geometric standard error = 1.10
Statistical Analysis 1: Comparison: Zongertinib Alone (Reference, R) vs Zongertinib+Carbamazepine (Test, T); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted geometric mean ratio (%) = 56.44, 90% CI 2-sided [45.11 to 70.60] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 37.9

3. Secondary Outcome: Area Under the Concentration-time Curve of Zongertinib in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of Zongertinib in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz).
  Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: hour * nanomole / liter (h*nmol/L)
Groups:
- Zongertinib (BI 1810631) Alone (Reference, R): In the reference treatment period (Period 1), participants were administered a single oral dose of 60 milligrams (mg) of Zongertinib in tablet form following an overnight fast of at least 10 hours, with 240 milliliters (mL) of water.
Arm/Group | Zongertinib (BI 1810631) Alone (Reference, R) | Zongertinib+Carbamazepine (Test, T)
Number analyzed (Participants) | 16 | 15
hour * nanomole / liter (h*nmol/L) | 12138.26 (NA) — Adjusted geometric standard error = 1.06 | 4430.05 (NA) — Adjusted geometric standard error = 1.06
Statistical Analysis 1: Comparison: Zongertinib (BI 1810631) Alone (Reference, R) vs Zongertinib+Carbamazepine (Test, T); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted geometric mean ratio (%) = 36.50, 90% CI 2-sided [31.91 to 41.74] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 22.3

ADVERSE EVENTS:
Time Frame: AE collected: Zongertinib : Up to 14 days after the first Zongertinib administration. Zongertinib + Carbamazepine loading: From Day -18 to Day -12 in Period 2, 6 days. Carbamazepine loading: Carbamazepine loading: From Day -12 to Day 1 in Period 2 (second administration on zongertinib), 12 days. Zongertinib + Carbamazepine: Up to 14 days after the second Zongertinib administration. All cause-mortality: up to 48 days
Description: Treated set (TS): The treated set includes all subjects who were treated with at least one dose of Zongertinib.
Groups:
- Zongertinib: Participants were administered a single dose of 60 milligrams (mg) of Zongertinib film-coated tablet orally on Day 1 of Visit 2 with 240 milliliters (mL) of water after an overnight fast of at least 10 hours.
- Zongertinib+Carbamazepine Loading: Participants took 200 mg of carbamazepine after dinner for 4 days, followed by 400 mg after dinner for 2 days.
- Carbamazepine Loading: Participants took 400 mg of carbamazepine after dinner for 5 days, followed by 600 mg after dinner for 7 days.
- Zongertinib+Carbamazepine: Participants took 600 mg of carbamazepine in the evening after dinner for 6 days. They also took a single dose of a 60 mg Zongertinib film-coated tablet in the morning on Day 1 of Visit 3, after an overnight fast of at least 10 hours.
Arm/Group | Zongertinib | Zongertinib+Carbamazepine Loading | Carbamazepine Loading | Zongertinib+Carbamazepine
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 3/16 | 7/15 | 11/15 | 5/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zongertinib (N=16) | Zongertinib+Carbamazepine Loading (N=15) | Carbamazepine Loading (N=15) | Zongertinib+Carbamazepine (N=15)
Constipation (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Faeces hard (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 3 | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Body temperature increased (Investigations) | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 1 | 0 | 0
Initial insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-09-14): https://cdn.clinicaltrials.gov/large-docs/64/NCT06028464/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-03): https://cdn.clinicaltrials.gov/large-docs/64/NCT06028464/SAP_001.pdf